CLINICAL TRIAL: NCT00113724
Title: A Phase I, Open-Label, Dose Escalation, Multi-Center Study of TPI 287 in Patients With Advanced Malignancies
Brief Title: Study of TPI 287 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortice Biosciences, Inc. (Industry)
Responsible Party: Tapestry Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPI 287-01
Expanded Access: Available
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2009-06-04 (Estimated); Status verified 2009-06

CONDITIONS: Neoplasms; Non-Hodgkin Lymphoma; Hodgkin Disease
Keywords: taxane; multi-drug resistance; mutant tubulin binding; Advanced malignancies; Hodgkin's or Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Neoplasms; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: TPI 287 Injection

SUMMARY:
Tapestry Pharmaceuticals, Inc. has developed a novel taxane analog, TPI 287. TPI 287 is synthetically manufactured from naturally occurring taxanes extracted from yew starting material. The synthesis involves modification to the taxane side chain to overcome multidrug resistance and to achieve mutant tubulin binding. This study will be a multi-center, dose escalation, sequential group, phase I study evaluating the intravenous administration of TPI 287, a novel third generation taxane.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the maximum tolerated dose of TPI 287 for phase II clinical trials.

The secondary objectives of the study are:

* To determine the safety of TPI 287
* To determine antitumor activity of TPI 287
* To determine the pharmacokinetic profile of TPI 287
* To determine the pharmacodynamic profile of TPI 287

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of malignancy
* Patients must have either:

  * advanced solid tumors that have recurred or progressed following standard therapy, or
  * Hodgkin's or non-Hodgkin's lymphoma that has recurred or progressed following standard therapy, have not had a previous bone marrow transplant, and are not eligible for a bone marrow transplant.
* Failed at least one previous therapeutic regimen and either no longer are candidates for standard therapy, have no standard therapy available, or choose not to pursue standard therapy.
* Ambulatory with ECOG 0 or 1, and a life expectancy of >3 months.
* Judged by the investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits.
* Have ability to read, understand and provide written informed consent for the initiation of any study related procedures or have a legal representative to perform this function.
* If female, must have a negative pregnancy test within 21 days of start of treatment.
* Agree to the use of an effective method of contraception during the study and for 90 days following the last dose of medication.
* Patients with prior radiation therapy for brain metastasis or primary brain tumors are acceptable.

Exclusion Criteria:

* Prior radiation therapy or chemotherapy within 4 weeks (6 weeks for prior nitrosoureas or mitomycin)
* Another active medical condition(s) or organ disease(s) that may either compromise patient safety or interfere with the safety and/or outcome evaluation of the study drug. While this exclusion is not limited to the following abnormalities, if any of the following laboratory abnormalities are present, the patient should be excluded:

  * WBC < 3000/uL;
  * Absolute neutrophil count < 1500/uL;
  * Platelets < 100,000/uL;
  * Total bilirubin > 1.5 x upper limit of normal;
  * ALT or AST > 3 x upper limit of normal if no liver metastases or >5 upper limit of normal in the presence of liver metastases;
  * Serum creatinine > 1.5 x upper limit of normal;
  * INR >2.0.
* Patient has clinically significant cardiac co-morbidities or pulmonary impairment
* Patient or physician plans concomitant chemotherapy, radiation therapy, hormonal and/or biological treatment for cancer including immunotherapy while on study. Of note, therapy with LHRH for prostate cancer is acceptable.
* Patient has been treated with any investigational drug, investigational biologic, or investigational therapeutic device within 30 days of initiating study treatment.
* Tumor appears to involve a major artery or vein.
* Prior or concurrent significant CNS disease including stroke, except for primary or secondary malignancies.
* Less than 4 weeks since prior major surgery
* Known positive for HIV, Hepatitis B or C
* Concurrent chronic use of aspirin (325 mg/day or more)
* Concurrent or recent (within 1 month) use of thrombolytic agents, or full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters) Of note, therapy with low-molecular weight heparin is acceptable as long as the INR<2.0.
* Uncontrolled hypertension
* Grade II-IV peripheral vascular disease within the past year
* Prior allergic reactions to compounds of similar chemical or biologic composition to TPI 287, paclitaxel or taxotere, Cremophor-EL-P, or other study agents
* Significant traumatic injury within the past 4 weeks
* Ongoing or active infection requiring parenteral antibiotics or with a fever >38.1°C within 3 days of the first scheduled day of dosing
* Other concurrent uncontrolled illness which may interfere with the ability of the patient to participate in the trial
* Patients who are inpatients
* Grade II-IV peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of TPI 287

SECONDARY OUTCOMES:
To determine the safety of TPI 287
To determine the antitumor activity of TPI 287
To determine the pharmacokinetic profile of TPI 287
To determine the pharmacodynamic profile of TPI 287

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Tapestry Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Georgetown University Medical Center/Lombardi Cancer Center, Washington D.C., District of Columbia
  - New York Medical College, Valhalla, New York